CLINICAL TRIAL: NCT00226070
Title: Cross-section Study Among Patients Waiting for or Already Undergoing THA Followed by a RCT
Brief Title: Rehabilitation to Patients Over 65 Years Undergoing THA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1301500110; 1999-2-20
Record Dates: First submitted 2005-09-23; First posted 2005-09-26 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Hip Arthroplasty
Keywords: selfrated health,; SF-36,; rehabilitation,; total hip replacement,; patients above 65
MeSH Terms: interventions — Interviews as Topic

INTERVENTIONS:
Procedure: interview and advising
Behavioral: 3 follow up interviews and personal advising
Procedure: interview SF-36 self rated health

SUMMARY:
Patients over 65 years do not have a self care ability the surgery benefits them.

The aim of this study is development of a rehabilitation program based on patients' self-rated health.

1. A cross section study including 600 patients
2. RCT including 160 patients

DETAILED DESCRIPTION:
Fase 1: 600 patients waiting for or already having received total hip-/knee-replacement participated in a questionnaire study using SF- 36. The aim was to document self-rated health among this population.

Fase 2: Results from the cross section study form the base for the RCT, where 160 patients over 65 years undergoing THR, 80 patients are in an intervention group and 80 patients in a control group. A nurse intervention program is tested, and results from the study will form the base for a structured rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:patients over 65 years undergoing total hip replacement

-

Exclusion Criteria:

* patients dropping out

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-01-02 (Actual); Primary Completion 2008-03-31 (Actual); Study Completion 2010-04-20 (Actual)

PRIMARY OUTCOMES:
Selfrated health among the population shows significant dysfunction among patients over 75 years, patient living alone and patients depended on help from others

SECONDARY OUTCOMES:
undergoing
we know next year

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Soballe, MD, Professor, Principal Investigator — Ortopaedic Center, Aarhus University Hospital, Aarhus Denmark; Kjeld Soballe, Principal Investigator — Department of Orthopaedics, Aarhus University Hospital, Tage Hansensgade 10, DK-8000 Aarhus C; Kjeld Soballe, MD,DR.Med.,Prof., Principal Investigator — Aarhus University Hospitak,Ortopaedic center, Aarhus Denmark
Locations (6):
- Denmark (6):
  - Aarhus University Hospital, Aarhus
  - Kjeld Soballe, Orthopaedic center, University of Aarhus, Aarhus
  - Kjeld Soballe, Orthopaedic Center, Aarhus
  - Orthopaedic Center, Aarhus
  - Ortopaedic center, Aarhus University, Aarhus
  - University of Aarhus, Faculty of Health Sciences, Orthopaedic center, Aarhus

REFERENCES:
- [Derived] Hordam B, Sabroe S, Pedersen PU, Mejdahl S, Soballe K. Nursing intervention by telephone interviews of patients aged over 65 years after total hip replacement improves health status: a randomised clinical trial. Scand J Caring Sci. 2010 Mar;24(1):94-100. doi: 10.1111/j.1471-6712.2009.00691.x. Epub 2009 Apr 28. PMID 19422632